CLINICAL TRIAL: NCT03597204
Title: Colorectal Cancer (CRC) Screening in Hong Kong: an Analysis on Acceptability, Compliance, Diagnostic Accuracy and Clinical Outcomes
Brief Title: Effectiveness of Fecal Immunnochemical Test and Colonoscopy Screening in Hong Kong
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Joseph JY SUNG, Professor of Medicine and Therapeutics, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CEHR
Record Dates: First submitted 2018-06-18; First posted 2018-07-24 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fecal immunochemical test (FIT) (Active Comparator): Annual fecal immunochemical test (FIT) for up to five years and follow-up colonoscopy was arranged for those with FIT positive result
  Interventions: Diagnostic Test: Fecal immunochemical test (FIT)
- Colonoscopy (Active Comparator): Subjects in the retrospective cohort were allowed to choose one-off colonoscopy for CRC screening
  Interventions: Diagnostic Test: Colonoscopy

INTERVENTIONS:
Diagnostic Test: Fecal immunochemical test (FIT) — Annual fecal immunochemical test (FIT) for up to five years and follow-up colonoscopy was arranged for those with FIT positive result
  Arms: Fecal immunochemical test (FIT)
Diagnostic Test: Colonoscopy — Subjects in the retrospective cohort were allowed to choose one-off colonoscopy for CRC screening
  Arms: Colonoscopy

SUMMARY:
Colorectal neoplasm in Asia is now increasingly common and is rising in an alarming manner in Hong Kong. Population-based screening for colorectal cancer (CRC) should be implemented. With the establishment of the CUHK JC Bowel Cancer Education Centre in 2008, about 10,000 asymptomatic subjects aged 50-70 years have completed screening by either faeca immunochemical test (FIT)or colonoscopy till December 2012. From 2013 onwards, the centre invites subjects aged 40-70 years with risk factors for CRC to undergo screening by FIT on a yearly basis. If FIT result is positive, according to local practice, they will be offered a routine colonoscopy as they will be treated as symptomatic. Currently, about 2,500 subjects have received CRC screening in this new project. There will be 2,500 subjects more to be recruited to this till 31 December 2017. The investigators would like to carry out a prospective cohort study of these 2,500 subjects and also retrospectively review the cohort of 12,500 subjects who received CRC screening in the CUHK JC Bowel Cancer Education Centre.

The present study aims to:

1. . Evaluate the knowledge, attitude, perception, practice, perceived obstacles and changes in choice of CRC screening among the screening participants;
2. . Assess the levels of compliance across time among those who joined the screening programme, according to different subject characteristics;
3. . Explore the diagnostic accuracy of faecal immunochemical tests among subjects with different characteristics;
4. . Evaluate the risk factors for colorectal neoplasia and if applicable, devise and validate a risk scoring system for prediction of neoplasia in different colon sites;
5. . Evaluate the association between bowel preparation, colonoscopy withdrawal time and adenoma detection rate among those who received colonoscopy;
6. . Validation of the existing risk scoring systems for colorectal neoplasia from the literature, based on findings from subjects who received colonoscopy.
7. . Explore potential associations among colorectal neoplasia detected in different colon sites.

DETAILED DESCRIPTION:
BACKGROUND

Colorectal neoplasm in Asia is not less common compared to that of the Western population and screening for colorectal cancer (CRC) should be implemented. In the Asia Pacific Consensus for Colorectal Cancer, Fecal Occult Blood Test (FOBT) was recommended as the preferred test in resource limited areas in Asia. Yet, the preference of Asian in the options for CRC screening might be different. In a recent study from Hong Kong, most subjects preferred to use colonoscopy instead of stool tests as the screening tool.

A study from Asia showed that fecal immunochemical test (FIT) might be preferred because it obviates the need for dietary control. Educating the public about different options available is an important method to change the health seeking behavior of subjects. The CUHK JC Bowel Cancer Education Centre was established in 2008 with full funding from the Hong Kong Jockey Club Charities Trust. About 10,000 subjects received CRC screening by either FIT or colonoscopy till 31 December 2012. From 2013 onwards, the centre invites subjects aged 40-70 years with risk factors for CRC to undergo screening by FIT on a yearly basis. If FIT result is positive, according to local practice, they will be offered a routine colonoscopy as they will be treated as symptomatic. Currently, a total of about 2,500 asymptomatic subjects have received CRC screening in this new project and the Centre will continue to recruit 2,500 subjects more till 31 December 2017.

To inform future screening policy for implementation of population-based screening, it is important to explore the different aspects of this community-based CRC screening programme which include various indicators of programmatic performance.

STUDY AIMS

1. Evaluate the knowledge, attitude, perception, practice, perceived obstacles and changes in choice of CRC screening among the screening participants;
2. Assess the levels of compliance across time among those who joined the screening programme, according to different subject characteristics;
3. Explore the diagnostic accuracy of faecal immunochemical tests among subjects with different characteristics;
4. Evaluate the risk factors for colorectal neoplasia and if applicable, devise and validate a risk scoring system for prediction of neoplasia in different colon sites;
5. Evaluate the association between bowel preparation, colonoscopy withdrawal time and adenoma detection rate among those who received colonoscopy;
6. Validation of the existing risk scoring systems for colorectal neoplasia from the literature, based on findings from subjects who received colonoscopy.
7. Explore potential associations among colorectal neoplasia detected in different colon sites.
8. Evaluate the long-term protective effect of FIT and colonoscopy on CRC incidence and mortality and all-cause mortality.

METHODOLOGY

Retrospective cohort Demographic data, health behavior information and clinical outcomes of subjects who received CRC screening in CUHK Bowel Cancer Education Centre from December 2008 to Sept 2015 will be retrospectively reviewed without consent and analyzed.

Prospective cohort

1. Study subjects will be invited to join the study via routine health talk of a CRC screening program organized by CUHK JC Bowel Cancer Education Centre
2. Each eligible subject completed a self-administered survey, which consists of sociodemographic information, family history of CRC for a first-degree relative, past medical history, and use of chronic medications. The completeness of questionnaires is checked afterwards. Trained volunteers assist survey completion for the relatively illiterate participants. The investigators used a quantitative FIT (OC Sensor). Participants received information on procedures for collecting the FIT samples at home, according to the manufacturer's instructions. They are requested to return their collection tubes containing faecal specimens to the centre 6 days within the stool collection. For those with negative FIT, they will be reminded to continue the FIT screening on a yearly basis till 2018. For those subjects with FIT positive findings, according to local practice, they will be offered a routine colonoscopy as they will be treated as symptomatic. Subjects who undergo colonoscopy may receive a phone-call follow up every year for the period of the study to monitor the clinical outcome of the subject. Subjects develop symptoms suggestive of colorectal neoplasm will be worked up by the original team of investigators.

Long-term Follow-up Follow-up with respect to long-term CRC incidence, CRC-related mortality and all-cause mortality will be conducted by matching participants' unique identifier to the Clinical Data Analysis and Reporting System (CDARS), Hospital Authority. A diagnosis of CRC will be defined as cancer in the colon or rectum, according to ICD-9 coding of 153.0-154.1 or 154.8. Follow-up time will be measured from the date of enrolment to the date of diagnosis of CRC, date of death (CRC-related or other cause), or the end of follow up (30 Nov 2023), whichever came first. The Kaplan-Meier (KM) estimator will be used to calculate the cumulative risks of CRC incidence, CRC-related mortality and all-cause mortality

ELIGIBILITY:
Inclusion Criteria:

Retrospective cohort

1. Subjects received CRC screening in CUHK JC Bowel Cancer Education Centre from 2008 up to 30 Sept 2015

Prospective cohort

1. Subjects aged 40-75 who were asymptomatic of CRC from CUHK JC Bowel Cancer Education Centre
2. Informed consent available
3. Identified as having risk factors for CRC (defined as having a Asia Pacific Colorectal Screening (APCS) score 4-7; the presence of diabetes; body mass index ≥25 kg/m2; or the presence of family history of CRC)

Exclusion Criteria:

1. Subject with any lower gastrointestinal (GI) symptoms (including lower GI bleeding, change in bowel habit, anemia and weight loss)
2. Prior history of colonic diseases that might increase the risk of colorectal cancer (including colorectal neoplasm, inflammatory bowel disease)
3. Examination of the colon (e.g. colonoscopy, barium enema or CT/MR of the colon) within the past 5 years
4. History of colorectal surgery in the past
5. Any contraindication for colonoscopy

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15000 (Actual)
Dates: Start 2015-10-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of subjects diagnosed colonic adenoma, advanced adenoma or cancer | Up to three years
  The diagnostic accuracy of faecal immunochemical test in the selected high risk individuals. The number of subjects diagnosed colonic adenoma, advanced adenoma or cancer will be divided by the total number of selected high risk subjects received fecal immunochemical test
Long-term CRC incidence and mortality and all-cause mortality | At least 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Joseph JY Sung, MD, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- CUHK Jockey Club Bowel Cancer Education Centre, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhu Z, Lam TYT, Tang RSY, Wong SH, Lui RNS, Ng SSM, Wong SYS, Sung JJY. Triglyceride-glucose index (TyG index) is associated with a higher risk of colorectal adenoma and multiple adenomas in asymptomatic subjects. PLoS One. 2024 Nov 7;19(11):e0310526. doi: 10.1371/journal.pone.0310526. eCollection 2024. PMID 39509387